CLINICAL TRIAL: NCT05079438
Title: A Multicenter Randomized Controlled Stage III Clinical Study of Dendrobium Huoshanense Suppository in Locally Advanced Rectal Cancer Patients Treated by Neoadjuvant Chemoradiotherapy
Brief Title: Dendrobium Huoshanense Suppository in Rectal Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, zhuji, Professor, Zhejiang Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CARTOnG-2103
Record Dates: First submitted 2021-10-01; First posted 2021-10-15 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: Locally Advanced Rectal Cancer
Keywords: Neoadjuvant Chemoradiotherapy; Dendrobium Huoshanense; irinotecan; capecitabine

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CRT with Dendrobium huoshanense Suppository (Experimental): Dendrobium huoshanense Suppository: 1.7g rectal administration per day for 5 weeks
  Concurrent Chemoradiotherapy:
  Radiation: 50Gy/25Fx; Capecitabine: 625mg/m2 bid Monday-Friday per week; Irinotecan: 80mg/m2 (UGT1A1*28 and *6: 6/6+GG) or 65mg/m2 (UGT1A1*28 and *6 ：6/7+GG or 6/6+GA) or 50mg/m2 （UGT1A1*28 and *6 ：7/7+GG or 6/6+AA or 6/7+GA）.
  Interventions: Drug: Dendrobium Huoshanense Suppository
- CRT with Placebo (No Intervention): Placebo: 1.7g rectal administration per day for 5 weeks
  Concurrent Chemoradiotherapy:
  Radiation: 50Gy/25Fx; Capecitabine: 625mg/m2 bid Monday-Friday per week; Irinotecan: 80mg/m2 (UGT1A1*28 and *6: 6/6+GG) or 65mg/m2 (UGT1A1*28 and *6 ：6/7+GG or 6/6+GA) or 50mg/m2 （UGT1A1*28 and *6 ：7/7+GG or 6/6+AA or 6/7+GA）.

INTERVENTIONS:
Drug: Dendrobium Huoshanense Suppository — 1.7g rectal administration per day for 5 weeks
  Arms: CRT with Dendrobium huoshanense Suppository

SUMMARY:
To evaluates the role of Dendrobium Huoshanense Suppository for radiation proctitis in locally advanced rectal cancer treated by capecitabine and irinotecan based neoadjuvant chemoradiation.

ELIGIBILITY:
Inclusion Criteria:

1. pathological confirmed rectum adenocarcinoma
2. clinical stage T3-4 and/or N+
3. the distance from anal verge less than 10 cm
4. without distance metastases
5. performance status score: 0~1
6. without previous anti-cancer therapy
7. able to follow the protocol during the study period
8. sign the inform consen

Exclusion Criteria:

1. Pregnant or breastfeeding women
2. Those with other history of malignant disease in the past 5 years, except for cured skin cancer and cervical carcinoma in situ
3. If there is an uncontrolled history of epilepsy, central nervous system disease or mental disorder, the investigator may determine that the clinical severity may hinder the signing of informed consent or affect the patient's oral medication compliance.
4. Clinically severe (ie, active) heart disease, such as symptomatic coronary heart disease, New York Heart Association (NYHA) class II or more severe congestive heart failure or severe arrhythmia requiring medication intervention (see appendix 12), or a history of myocardial infarction in the last 12 months
5. Organ transplantation requires immunosuppressive therapy Severe uncontrolled recurrent infections, or other serious uncontrolled concomitant diseases
6. Subject blood routine and biochemical indicators do not meet the following criteria: hemoglobin ≥ 90g / L; absolute neutrophil count (ANC) ≥ 1.5 × 109 / L; Alanine transaminase (ALT), aspartate aminotransferase (AST) ≤ 2.5 times the upper limit of normal; alkaline phosphatase (ALP) ≤2.5 times the normal upper limit; serum total bilirubin <1.5 times the normal upper limit; serum creatinine <1 times the normal upper limit; serum albumin ≥ 30g / L
7. Anyone who is allergic to any research medication
8. DPD deficiency

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2021-09-07 (Actual); Primary Completion 2023-07-30 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
≥Grade 2 proctitis | During chemoradiotherapy

CONTACTS AND LOCATIONS:
Locations (1):
- Ji Zhu, Hangzhou, Zhejiang, China